CLINICAL TRIAL: NCT04947917
Title: Axillary Lymph Node Tattoo Marking Versus Biopsy Marker and Radioseed Tagging in Patients With Known Primary Breast Cancer
Brief Title: Axillary Lymph Node Tattoo Marking Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional standard of care regarding axillary management changed. Decision was made to close the study early.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Leah H Portnow, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-754
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Lymph Node Metastases
Keywords: Breast Cancer; Lymph Node Metastases
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymph Node SpotTM Tattoo (Experimental): Spot™ ink tattooing will be administered once prior to surgery.
  Initial test set of participants with previous sampled lymph nodes positive for metastasis will have SpotTM ink administered at time of standard of care pre-surgery radioseed localization.
  A feasibility set of participants will have SpotTM ink administered at time standard of care lymph nodes sampling.
  Interventions: Procedure: SpotTM Tattoo Ink

INTERVENTIONS:
Procedure: SpotTM Tattoo Ink — Ink injection

SUMMARY:
This research study investigates if SpotTM ink can help breast surgeons retrieve sampled lymph node as well as or better than the standard clip and radioseed guidance methods.

The names of the novel study intervention involved in this study is:

* SpotTM ink tattooing

The names of the standard of care study interventions involved in this study are:

* Core needle biopsy and/or fine needle aspiration
* Surgical Removal of the Lymph Nodes via clip and radioseed guidance

DETAILED DESCRIPTION:
This research study is a Feasibility Study, in which investigators are examining SpotTM ink to find out if retrieval rates of the inked lymph node at surgery are as good as or better than the standard of care, which is to clip and then radioseed-label the positive axillary lymph node.

This research study involves placement of SpotTM ink on the surface of the lymph node at the time of sampling. As per standard of care, if the lymph node is positive for malignant cells, the surgeon will remove the lymph node at the time of surgical excision. The lymph node tissue will then be evaluated by the pathologist.

The U.S. Food and Drug Administration (FDA) has approved SpotTM ink for use in the large intestine to mark colon polyps. The FDA has not approved SpotTM ink for use in axillary lymph nodes. However, SpotTM ink has been used in axillary lymph nodes by other institutions in smaller studies similar to this one with success in retrieving the lymph node after surgery.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will be in this research study until surgical removal of their breast cancer and lymph nodes after their tattoo ink placement.

ELIGIBILITY:
Inclusion Criteria:

Any patient presenting with a new diagnosis of breast cancer or with imaging findings highly suspicious for breast cancer (BI-RADS® 4C and 5) and suspicious axillary lymph node(s) is potentially eligible. Inclusion criteria are those eligible patients who have axillary lymph node(s) that are suspicious by imaging. Evaluation of the axilla with US will be performed when clinically warranted, with lymph node sampling recommended by the radiologist based on morphologically abnormal features.

* Age 18 years. Because no dosing or adverse event data are currently available on the use of Spot™ ink in participants <18 years of age, children are excluded from this study.

Patients must be able to undergo breast imaging and surgical procedures, and therefore have a ECOG performance status ≤2 (Karnofsky ≥60%).

* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Women who are pregnant or lactating are eligible as Spot™ ink is placed focally in the axillary lymph node and breast tissues.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Exclusion criteria includes patients who have upper body or ipsilateral arm tattoos, as that ink may already be present in regional nodes and may confound visibility of Spot™ ink [19]. If NAC has already been initiated and the lymph node is no longer visualized, tattooing will not be performed, and that patient will also be excluded.

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Spot™ ink.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Retrieval Rate | Enrollment to completion of surgery up to 1 year
  The primary endpoint is feasibility. Feasibility will be defined by the successful intra-operative rate of retrieval of the lymph nodes tagged by SpotTM ink versus the clip and radioseed.

SECONDARY OUTCOMES:
Cost savings | Enrollment to completion of surgery up to 1 year
  Extrapolated by calculating cost-savings of Spot™ ink vs. clipped and radioseed-labelling lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Leah H Portnow, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation